CLINICAL TRIAL: NCT00718666
Title: Long Term Antibody Persistence Study of GSK Biologicals' Meningococcal Vaccine GSK 134612 Administered as 1 or 2 Doses to Healthy Toddlers at 9-12 Months of Age and as a Booster Dose at 5 Years Post-primary Vaccination
Brief Title: The Long-term Antibody Persistence of GSK Biologicals' Meningococcal Vaccine GSK134612 in Healthy Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112021; 2012-002719-24 (EudraCT Number)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Infections, Meningococcal
Keywords: Safety; Vaccines, conjugate; Immunogenicity; Meningococcal vaccine; Booster vaccination; Primary vaccination; Neisseria meningitides; Toddlers; Humans; Meningococcal disease
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal

ARMS (3):
- Group A (Experimental): Subjects who were previously vaccinated with one dose of GSK134612 at 12 months of age.
  Interventions: Biological: Meningococcal vaccine GSK134612
- Group B (Experimental): Subjects who were previously vaccinated with two doses of GSK134612, one each at 9 and 12 months of age.
  Interventions: Biological: Meningococcal vaccine GSK134612
- Group C (Experimental): Subjects aged 5-6 years not previously administered meningococcal vaccine.
  Interventions: Biological: Meningococcal vaccine GSK134612

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One dose, as intramuscular injection

SUMMARY:
In this study, the concentration of antibody to the vaccine one year, three and five years after vaccination in subjects who were vaccinated with GSK Biologicals' meningococcal vaccine GSK134612 in a previous study (whose objectives & outcome measures are presented in a separate protocol posting with NCT number =00471081) will be evaluated. The safety and immune response of a booster dose of vaccine GSK134612 administered at 5 years post-primary vaccination will also be evaluated. In addition, the immune response to a dose of vaccine GSK134612 administered to age-matched controls not previously given a meningococcal vaccine will be evaluated.

This protocol posting has been updated further to protocol amendment 2, dated 28 october 2010. The sections impacted are summary, study design, outcome measures, intervention, and eligibility criteria.

DETAILED DESCRIPTION:
GSK Biologicals has developed a meningococcal conjugate vaccine (GSK134612). This candidate vaccine has been shown to be well tolerated and immunogenic in toddlers.

The purpose of this study is to evaluate the antibody persistence at approximately 1 year, 3 years and 5 years post-administration of one dose or two doses of GlaxoSmithKline (GSK) Biologicals' meningococcal vaccine GSK134612 when given to healthy toddlers 9-12 months of age. To evaluate, the safety and immunogenicity of a booster dose of GSK134612 administered to all eligible subjects at 5 years after the primary vaccination. To evaluate the safety and immunogenicity in a new group of subjects aged 5-6 years (naive control group) who will receive a single dose of vaccine GSK134612.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria for the persistence phase of the study entry:

* A male or female toddler who was vaccinated 1, 3 or 5 years ago with the last dose of MenACWY-TT in study with NCT number=00471081.
* Written informed consent obtained from parents/guardian of the subject.
* Healthy subjects as established by medical history before entering into the study.
* Having completed the active phase of the vaccination study with NCT number=00471081 (i.e., not withdrawn, had received all planned doses of study vaccines, provided a post-vaccination blood sample after the final dose).

All subjects must meet the following criteria prior to receiving the booster vaccination:

* Written informed consent obtained from parents/guardian of the subject.
* Subjects who can and will comply with the requirements of the protocol.
* Subjects who provide a blood sample 5 years after last vaccination in study with NCT number=00471081.

All subjects must satisfy the following criteria prior to enrollment in the naïve control group:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female between, and including, 5-6 years of age at the time of the vaccination.
* Written informed consent obtained from parents/guardian of the subject.
* Healthy subjects as established by medical history and history-directed physical examination before entering into the study.

Exclusion Criteria:

Exclusion criteria for persistence study entry

* Use of any investigational or non-registered product (drug or vaccine) within 30 days of each persistence timepoint.
* Vaccination with meningococcal polysaccharide or conjugate vaccine of serogroup A, B, C, W-135, and/or Y outside of study with NCT number=00471081.
* History of any meningococcal disease due to serogroup A, B, C, W-135, or Y.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition based on medical history and physical examination (no laboratory testing is required).
* Administration of immunoglobulins and/or any blood products within the three months preceding each persistence timepoint.
* Concurrently participating in another clinical study within 30 days of each persistence timepoint, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* Subjects withdrew consent to be contacted for follow-up studies.

Exclusion criteria for primary (naive control)/booster vaccination at year 5 study entry (to be checked at Year 5)

* Child in care.
* Subjects who were enrolled in the Kaiser Healthcare system in study with NCT number=00471081, but are no longer enrolled.
* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the primary (naive control)/booster vaccination, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the primary (naive control)/booster vaccination. (For corticosteroids, this will mean prednisone, or equivalent, >= 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Vaccination with meningococcal polysaccharide or conjugate vaccine outside of study with NCT number=00471081.
* History of any meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history (no laboratory testing is required).
* Administration of immunoglobulins and/or any blood products within the three months preceding the primary (naive control)/booster vaccination or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* Subjects withdrew consent to be contacted for follow-up studies.
* Hypersensitivity to latex.
* Previous administration or planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days of the study vaccination (primary vaccination for the naïve control group and booster vaccination for subjects primed in Study with NCT number = 00471081) and ending 30 days after with the exception of any licensed inactivated influenza vaccine (live attenuated influenza vaccine is not allowed).
* Previous administration or planned administration of tetanus or any tetanus containing vaccine during the period starting from 30 days of the study vaccination and ending 30 days after.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease at the time of vaccination. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., temperature by any method < 99.5°F (37.5°C).

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 387 (Actual)
Dates: Start 2008-10-20 (Actual); Primary Completion 2013-11-13 (Actual); Study Completion 2014-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (13):
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vacaville, California
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Westminster, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Amarillo, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Klein NP, Baine Y, Bianco V, Lestrate PR, Naz A, Blatter M, Friedland LR, Miller JM. One or two doses of quadrivalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine is immunogenic in 9- to 12-month-old children. Pediatr Infect Dis J. 2013 Jul;32(7):760-7. doi: 10.1097/INF.0b013e31828693c5. PMID 23348814
- [Background] Klein NP, Baine Y, Kolhe D, Baccarini CI, Miller JM, Van der Wielen M. Five-year Antibody Persistence and Booster Response After 1 or 2 Doses of Meningococcal A, C, W and Y Tetanus Toxoid Conjugate Vaccine in Healthy Children. Pediatr Infect Dis J. 2016 Jun;35(6):662-72. doi: 10.1097/INF.0000000000001123. PMID 26928521
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not all study participants returned in time for every study visit, but they were allowed to continue the study nonetheless. The number of participants who started each study period depends on the actual rate of return of the subjects.
Pre-assignment Details: Out of 387 subjects originally enrolled in the study, only 248 subjects received vaccination.
Groups:
- Nimenrix 1 Group: Subjects who received 1 dose of Nimenrix vaccine at 12 months of age.
- Nimenrix 2 Group: Subjects who were previously vaccinated with two doses of Nimenrix, one each at 9 and 12 months of age.
- Nimenrix Naive Group: Vaccine-naive subjects aged 5-6 years were enrolled to receive Nimenrix vaccine as primary vaccination at Year 5.
Period: Persistence Phase Year 1
Arm/Group | Nimenrix 1 Group | Nimenrix 2 Group | Nimenrix Naive Group
Started | 118 | 130 | 0
Completed | 118 | 130 | 0 (Subjects enrolled to receive Nimenrix vaccine as primary vaccination only at Booster Phase-Year 5.)
Not Completed | 0 | 0 | 0
Period: Persistence Phase Year 3
Arm/Group | Nimenrix 1 Group | Nimenrix 2 Group | Nimenrix Naive Group
Started | 98 | 104 | 0
Completed | 98 | 104 | 0 (Subjects enrolled to receive Nimenrix vaccine as primary vaccination only at Booster Phase-Year 5.)
Not Completed | 0 | 0 | 0
Period: Persistence Phase Year 5
Arm/Group | Nimenrix 1 Group | Nimenrix 2 Group | Nimenrix Naive Group
Started | 70 | 82 | 0
Completed | 70 | 82 | 0 (Subjects enrolled to receive Nimenrix vaccine as primary vaccination only at Booster Phase-Year 5.)
Not Completed | 0 | 0 | 0
Period: Booster Phase Year 5
Arm/Group | Nimenrix 1 Group | Nimenrix 2 Group | Nimenrix Naive Group
Started | 38 | 46 | 100
Completed | 36 | 46 | 94
Not Completed | 2 | 0 | 6
Not completed — No active participation request | 0 | 0 | 1
Not completed — Declined v-4 serology | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Period for Nimenrix 1 Group and Nimenrix 2 Group is considered Year 1 and Baseline Period for Nimenrix Naive Group is considered Year 5.
Groups:
- Nimenrix 1 Group Y1: Subjects from Year 1 Period who received 1 dose on Nimenrix vaccine at 12 months of age.
- Nimenrix 2 Group Y1: Subjects from Year 1 Period who were previously vaccinated with two doses of Nimenrix, one each at 9 and 12 months of age.
- Total: Total of all reporting groups
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1 | Nimenrix Naive Group | Total
Number analyzed (Participants) | 118 | 130 | 100 | 348
Age, Continuous [Mean (Standard Deviation); unit: Months] | 24.5 (0.97) | 24.6 (1.00) | 69.2 (6.6) | 37.38 (20.56)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 56 | 66 | 44 | 166
  Male | 62 | 64 | 56 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 7 | 7 | 23 | 37
  Geographic ancestry: American Indian or Alaskan Native | 9 | 16 | 10 | 35
  Geographic ancestry: Asian-Central/South Asian heritage | 3 | 4 | 1 | 8
  Geographic ancestry: Asian-East Asian heritage | 2 | 0 | 0 | 2
  Geographic ancestry: Asian-South East Asian heritage | 7 | 8 | 3 | 18
  Geographic ancestry: Native Hawaiian or other Pacific Islander | 1 | 2 | 3 | 6
  Geographic ancestry: White-Arabic/North African heritage | 1 | 0 | 1 | 2
  Geographic ancestry: White-Caucasian/European heritage | 72 | 67 | 46 | 185
  Geographic ancestry: Other | 16 | 26 | 13 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay (Using Human Complement) (hSBA) Titers ≥ the Cut-off
Description: hSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off value assessed was greater than or equal to ( ≥) 1:8.
Time Frame: At Year 1 (12 months post primary vaccination)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence Year 1, which included all evaluable subjects who were eligible in the primary study 109375, who complied with the protocol requirements and for whom assay results for at least 1 tested antigen were available at the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1
Number analyzed (Participants) | 110 | 120
Participants
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 102 | 108
  hSBA-MenA, ≥ 1:8 | 21 | 28
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 104 | 113
  hSBA-MenC, ≥ 1:8 | 91 | 103
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 104 | 112
  hSBA-MenW-135, ≥ 1:8 | 93 | 111
  hSBA-MenY, ≥ 1:8 | 88 | 111

2. Primary Outcome: Number of Subjects With Serum Bactericidal Assay (Using Human Complement) (hSBA) Titers ≥ the Cut-off
Description: hSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off value assessed was ≥ 1:8.
Time Frame: At Year 3 (36 months post primnary vaccination)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence Year 3, which included all evaluable subjects who were eligible in the primary study 109375, who complied with the protocol requirements and for whom assay results for at least 1 tested antigen were available at the considered time point.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 1 Group Y3: Subjects from Year 3 Period who received 1 dose on Nimenrix vaccine at 12 months of age.
- Nimenrix 2 Group Y3: Subjects from Year 3 Period who were previously vaccinated with two doses of Nimenrix, one each at 9 and 12 months of age.
Arm/Group | Nimenrix 1 Group Y3 | Nimenrix 2 Group Y3
Number analyzed (Participants) | 86 | 97
Participants
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 82 | 96
  hSBA-MenA, ≥ 1:8 | 14 | 16
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 81 | 94
  hSBA-MenC, ≥ 1:8 | 57 | 68
  hSBA-MenW-135, ≥ 1:8 | 54 | 82
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 85 | 95
  hSBA-MenY, ≥ 1:8 | 53 | 59

3. Primary Outcome: Number of Subjects With Serum Bactericidal Assay (Using Human Complement) (hSBA) Titers ≥ the Cut-off Values
Description: as for outcome 2
Time Frame: At Year 5 (60 months post primary vaccination)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence Year 5, which included all evaluable subjects who were eligible in the primary study 109375, who complied with the protocol requirements and for whom assay results for at least 1 tested antigen were available at the considered time point.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 1 Group Y5: Subjects from Year 5 Period who received 1 dose on Nimenrix vaccine at 12 months of age.
- Nimenrix 2 Group Y5: Subjects from Year 5 period who were previously vaccinated with two doses of Nimenrix, one each at 9 and 12 months of age.
Arm/Group | Nimenrix 1 Group Y5 | Nimenrix 2 Group Y5
Number analyzed (Participants) | 63 | 72
Participants
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 63 | 71
  hSBA-MenA, ≥ 1:8 | 20 | 27
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 60 | 71
  hSBA-MenC, ≥ 1:8 | 45 | 53
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 61 | 72
  hSBA-MenW-135, ≥ 1:8 | 40 | 62
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 50 | 63
  hSBA-MenY, ≥ 1:8 | 32 | 49

4. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY Titers ≥ the Cut-off Values
Description: hSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off value assessed was ≥ 1:4.
Time Frame: At Year 1 (12 months post vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1
Number analyzed (Participants) | 110 | 120
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 102 | 108
  hSBA-MenA, ≥ 1:4 | 23 | 29
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 104 | 113
  hSBA-MenC, ≥ 1:4 | 91 | 103
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 104 | 112
  hSBA-MenW-135, ≥ 1:4 | 93 | 111
  hSBA-MenY, ≥ 1:4 | 89 | 111

5. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY Titers ≥ the Cut-off Values
Description: as for outcome 4
Time Frame: At Year 3 (36 months post primary vaccination)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y3 | Nimenrix 2 Group Y3
Number analyzed (Participants) | 86 | 97
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 82 | 96
  hSBA-MenA, ≥ 1:4 | 14 | 19
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 81 | 94
  hSBA-MenC, ≥ 1:4 | 59 | 69
  hSBA-MenW-135, ≥ 1:4 | 54 | 82
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 85 | 95
  hSBA-MenY, ≥ 1:4 | 53 | 59

6. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY Titers ≥ the Cut-off Values
Description: as for outcome 4
Time Frame: At Year 5 (60 months post primary vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y5 | Nimenrix 2 Group Y5
Number analyzed (Participants) | 63 | 72
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 63 | 71
  hSBA-MenA, ≥ 1:4 | 20 | 27
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 60 | 71
  hSBA-MenC, ≥ 1:4 | 47 | 56
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 61 | 72
  hSBA-MenW-135, ≥ 1:4 | 40 | 62
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 50 | 63
  hSBA-MenY, ≥ 1:4 | 32 | 49

7. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) for the serogroups hSBA-MenA, hSBA-MenC, hSBAMenW-135, and hSBA-MenY respectively, calculated on all subjects.
Time Frame: At Year 1 (12 months post primary vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1
Number analyzed (Participants) | 110 | 120
Titres
  hSBA-MenA: number analyzed (Participants) | 102 | 108
  hSBA-MenA | 3.7 [2.9 to 4.8] | 4.1 [3.2 to 5.2]
  hSBA-MenC: number analyzed (Participants) | 104 | 113
  hSBA-MenC | 70.5 [50.4 to 98.5] | 72.4 [53.3 to 98.4]
  hSBA-MenW-135: number analyzed (Participants) | 104 | 112
  hSBA-MenW-135 | 127.9 [87.3 to 187.3] | 204.6 [163.6 to 255.9]
  hSBA-MenY | 55.6 [38.1 to 81.1] | 86.2 [65.8 to 112.9]

8. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY Antibody Titers
Description: as for outcome 7
Time Frame: At Year 3 (36 months post primary vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix 1 Group Y3 | Nimenrix 2 Group Y3
Number analyzed (Participants) | 86 | 97
Titres
  hSBA-MenA: number analyzed (Participants) | 82 | 96
  hSBA-MenA | 3.5 [2.6 to 4.6] | 3.4 [2.7 to 4.3]
  hSBA-MenC: number analyzed (Participants) | 81 | 94
  hSBA-MenC | 31.2 [18.9 to 51.6] | 29.8 [18.9 to 47]
  hSBA-MenW-135 | 29 [18 to 46.9] | 63.9 [44 to 92.8]
  hSBA-MenY: number analyzed (Participants) | 85 | 95
  hSBA-MenY | 22 [14 to 34.5] | 20.5 [13.6 to 30.8]

9. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-MenY Antibody Titers
Description: as for outcome 7
Time Frame: At Year 5 (60 months post primary vaccination)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix 1 Group Y5 | Nimenrix 2 Group Y5
Number analyzed (Participants) | 63 | 72
Titres
  hSBA-MenA: number analyzed (Participants) | 63 | 71
  hSBA-MenA | 4.6 [3.3 to 6.3] | 6.6 [4.5 to 9.8]
  hSBA-MenC: number analyzed (Participants) | 60 | 71
  hSBA-MenC | 40.7 [22.7 to 73.1] | 38.2 [22.5 to 64.9]
  hSBA-MenW-135: number analyzed (Participants) | 61 | 72
  hSBA-MenW-135 | 24.2 [14.4 to 40.7] | 53.7 [35.8 to 80.4]
  hSBA-MenY: number analyzed (Participants) | 50 | 63
  hSBA-MenY | 26 [14.1 to 47.8] | 37.9 [24.3 to 59.2]

10. Secondary Outcome: Number of Subjects With Titers ≥ the Cut-off for Meningococcal Polysaccharides A , C, W-135 and Y Serum Bactericidal Antibodies, Using Baby Rabbit Complement for Assay
Description: rSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off value assessed were ≥ 1:8 and 1:128. The analysis was performed by GSK Biologicals' laboratory assay.
Time Frame: At Year 1 (12 months post primary vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1
Number analyzed (Participants) | 101 | 114
Participants
  rSBA-MenA, ≥ 1:8: number analyzed (Participants) | 95 | 104
  rSBA-MenA, ≥ 1:8 | 90 | 101
  rSBA-MenA, ≥ 1:128: number analyzed (Participants) | 95 | 104
  rSBA-MenA, ≥ 1:128 | 71 | 80
  rSBA-MenC, ≥ 1:8: number analyzed (Participants) | 95 | 112
  rSBA-MenC, ≥ 1:8 | 83 | 96
  rSBA-MenC, ≥ 1:128: number analyzed (Participants) | 95 | 112
  rSBA-MenC, ≥ 1:128 | 46 | 54
  rSBA-MenW-135, ≥ 1:8 | 97 | 114
  rSBA-MenW-135, ≥ 1:128 | 82 | 89
  rSBA-MenY, ≥ 1:8: number analyzed (Participants) | 101 | 113
  rSBA-MenY, ≥ 1:8 | 96 | 113
  rSBA-MenY, ≥ 1:128: number analyzed (Participants) | 101 | 113
  rSBA-MenY, ≥ 1:128 | 85 | 100

11. Secondary Outcome: Number of Subjects With Titers ≥ the Cut-off, for MenA , MenC, MenW-135 and MenY Serum Bactericidal Antibodies, Using Baby Rabbit Complement
Description: as for outcome 10
Time Frame: At Year 3 (36 months post primary vaccination)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y3 | Nimenrix 2 Group Y3
Number analyzed (Participants) | 73 | 89
Participants
  rSBA-MenA, ≥ 1:8: number analyzed (Participants) | 69 | 84
  rSBA-MenA, ≥ 1:8 | 65 | 82
  rSBA-MenA, ≥ 1:128: number analyzed (Participants) | 69 | 84
  rSBA-MenA, ≥ 1:128 | 51 | 65
  rSBA-MenC, ≥ 1:8: number analyzed (Participants) | 68 | 89
  rSBA-MenC, ≥ 1:8 | 60 | 75
  rSBA-MenC, ≥ 1:128: number analyzed (Participants) | 68 | 89
  rSBA-MenC, ≥ 1:128 | 32 | 40
  rSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 72 | 88
  rSBA-MenW-135, ≥ 1:8 | 68 | 88
  rSBA-MenW-135, ≥ 1:128: number analyzed (Participants) | 72 | 88
  rSBA-MenW-135, ≥ 1:128 | 56 | 69
  rSBA-MenY, ≥ 1:8 | 69 | 89
  rSBA-MenY, ≥ 1:128 | 62 | 78

12. Secondary Outcome: Number of Subjects With Titers ≥ the Cut-off for Meningococcal Polysaccharides A , C, W-135 and Y Serum Bactericidal Antibodies, Using Baby Rabbit Complement for Assay
Description: rSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off values assessed were ≥ 1:8 and 1:128. Titers were determined by Public Health England (PHE) laboratory assay.
Time Frame: At Year 3 (36 months post primary vaccination)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y3 | Nimenrix 2 Group Y3
Number analyzed (Participants) | 83 | 98
Participants
  rSBA-MenA, ≥ 1:8: number analyzed (Participants) | 83 | 97
  rSBA-MenA, ≥ 1:8 | 38 | 44
  rSBA-MenA, ≥ 1:128: number analyzed (Participants) | 83 | 97
  rSBA-MenA, ≥ 1:128 | 23 | 24
  rSBA-MenC, ≥ 1:8: number analyzed (Participants) | 83 | 97
  rSBA-MenC, ≥ 1:8 | 27 | 30
  rSBA-MenC, ≥ 1:128: number analyzed (Participants) | 83 | 97
  rSBA-MenC, ≥ 1:128 | 18 | 15
  rSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 83 | 95
  rSBA-MenW-135, ≥ 1:8 | 36 | 35
  rSBA-MenW-135, ≥ 1:128: number analyzed (Participants) | 83 | 95
  rSBA-MenW-135, ≥ 1:128 | 24 | 23
  rSBA-MenY, ≥ 1:8 | 39 | 45
  rSBA-MenY, ≥ 1:128 | 21 | 24

13. Secondary Outcome: Number of Subjects With Titers ≥ the Cut-off, for Meningococcal Polysaccharides A , C, W-135 and Y Serum Bactericidal Antibodies, Using Baby Rabbit Complement for Assay
Description: rSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off values assessed were ≥ 1:8 and 1:128. The analysis was performed by GSK Biologicals' laboratory assay.
Time Frame: At Year 5 (60 months post-primary vacccination).
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y5 | Nimenrix 2 Group Y5
Number analyzed (Participants) | 53 | 64
Participants
  rSBA-MenA, ≥ 1:8: number analyzed (Participants) | 51 | 59
  rSBA-MenA, ≥ 1:8 | 51 | 57
  rSBA-MenA, ≥ 1:128: number analyzed (Participants) | 51 | 59
  rSBA-MenA, ≥ 1:128 | 38 | 49
  rSBA-MenC, ≥ 1:8: number analyzed (Participants) | 51 | 63
  rSBA-MenC, ≥ 1:8 | 43 | 53
  rSBA-MenC, ≥ 1:128: number analyzed (Participants) | 51 | 63
  rSBA-MenC, ≥ 1:128 | 23 | 31
  rSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 52 | 64
  rSBA-MenW-135, ≥ 1:8 | 51 | 64
  rSBA-MenW-135,≥ 1:128: number analyzed (Participants) | 52 | 64
  rSBA-MenW-135,≥ 1:128 | 41 | 53
  rSBA-MenY, ≥ 1:8 | 50 | 64
  rSBA-MenY, ≥ 1:128 | 43 | 58

14. Secondary Outcome: Number of Subjects With Titers ≥ the Cut-off for Men-A , Men-C, Men-W-135 and Men-Y Serum Bactericidal Antibodies, Using Baby Rabbit Complement for Assay
Description: rSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off values assessed were ≥ 1:8 and 1:128 determined by Public Health England (PHE) laboratory assay.
Time Frame: At Year 5 (60 months post-primary vacccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y5 | Nimenrix 2 Group Y5
Number analyzed (Participants) | 62 | 72
Participants
  rSBA-MenA, ≥ 1:8: number analyzed (Participants) | 61 | 72
  rSBA-MenA, ≥ 1:8 | 38 | 42
  rSBA-MenA, ≥ 1:128: number analyzed (Participants) | 61 | 72
  rSBA-MenA, ≥ 1:128 | 22 | 26
  rSBA-MenC, ≥ 1:8: number analyzed (Participants) | 62 | 71
  rSBA-MenC, ≥ 1:8 | 29 | 29
  rSBA-MenC, ≥ 1:128: number analyzed (Participants) | 62 | 71
  rSBA-MenC, ≥ 1:128 | 16 | 19
  rSBA-MenW-135, ≥ 1:8 | 15 | 22
  rSBA-MenW-135, ≥ 1:128 | 9 | 14
  rSBA-MenY, ≥ 1:8: number analyzed (Participants) | 61 | 72
  rSBA-MenY, ≥ 1:8 | 33 | 36
  rSBA-MenY, ≥ 1:128: number analyzed (Participants) | 61 | 72
  rSBA-MenY, ≥ 1:128 | 23 | 26

15. Secondary Outcome: rSBA Antibody Titers
Description: Titers were given as geometric mean titers (GMTs) for the serogroups rSBA-MenA, rSBA-MenC, rSBAMenW-135, and rSBA-MenY respectively, as performed by GSK Biologicals' laboratory assay.
Time Frame: At Year 1 (12 months post primary vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1
Number analyzed (Participants) | 101 | 114
Titers
  rSBA-MenA: number analyzed (Participants) | 95 | 104
  rSBA-MenA | 259.7 [191.4 to 352.3] | 237.2 [187 to 301]
  rSBA-MenC: number analyzed (Participants) | 95 | 112
  rSBA-MenC | 94.1 [67.1 to 131.9] | 90.3 [65.5 to 124.4]
  rSBA-MenW-135 | 385.2 [286.4 to 518.1] | 345.3 [280.1 to 425.8]
  rSBA-MenY: number analyzed (Participants) | 101 | 113
  rSBA-MenY | 364.5 [273.7 to 485.4] | 342.2 [284.5 to 411.8]

16. Secondary Outcome: rSBA Antibody Titers.
Description: Titers are given as geometric mean titers (GMTs) for the serogroups rSBA-MenA, rSBA-MenC, rSBAMenW-135, and rSBA-MenY respectively, as performed by GSK Biologicals' laboratory assay.
Time Frame: At Year 3 (36 months post-primary vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Group Y3 | Nimenrix 2 Group Y3
Number analyzed (Participants) | 73 | 89
Titers
  rSBA-MenA: number analyzed (Participants) | 69 | 84
  rSBA-MenA | 247.9 [173.8 to 353.7] | 241.8 [185.6 to 315]
  rSBA-MenC: number analyzed (Participants) | 68 | 89
  rSBA-MenC | 87 [59.3 to 127.8] | 76.4 [53.5 to 109]
  rSBA-MenW-135: number analyzed (Participants) | 72 | 88
  rSBA-MenW-135 | 353.3 [240 to 520.1] | 358 [282.8 to 453.3]
  rSBA-MenY | 360.5 [253.4 to 512.9] | 341.4 [276.9 to 421.1]

17. Secondary Outcome: rSBA Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) for the serogroups rSBA-MenA, rSBA-MenC, rSBA-MenW-135, and rSBA-MenY respectively. Titers were determined by Public Health England (PHE) laboratory assay.
Time Frame: At Year 3 (36 months following primary vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Nimenrix 1 Group Y3: Subjects who received 1 dose on Nimenrix vaccine at 12 months of age.
- Nimenrix 2 Group Y3: Subjects who were previously vaccinated with two doses of Nimenrix, one each at 9 and 12 months of age.
Arm/Group | Nimenrix 1 Group Y3 | Nimenrix 2 Group Y3
Number analyzed (Participants) | 83 | 98
Titers
  rSBA-MenA: number analyzed (Participants) | 83 | 97
  rSBA-MenA | 18.4 [12 to 28.3] | 16.6 [11.3 to 24.3]
  rSBA-MenC: number analyzed (Participants) | 83 | 97
  rSBA-MenC | 13.2 [8.6 to 20.2] | 10.6 [7.4 to 15]
  rSBA-MenW-135: number analyzed (Participants) | 83 | 95
  rSBA-MenW-135 | 19.4 [12.3 to 30.6] | 14.6 [9.7 to 21.8]
  rSBA-MenY | 19.6 [12.7 to 30.1] | 16.7 [11.5 to 24.3]

18. Secondary Outcome: rSBA Antibody Titers
Description: Titers are given as geometric mean titers (GMTs), calculated on all subjects for the serogroups rSBA-MenA, rSBA-MenC, rSBAMenW-135, and rSBA-MenY respectively by GSK Biologicals' laboratory assay.
Time Frame: At Year 5 (60 months post-primary vacccination)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Group Y5 | Nimenrix 2 Group Y5
Number analyzed (Participants) | 53 | 64
Titers
  rSBA-MenA: number analyzed (Participants) | 51 | 59
  rSBA-MenA | 311.6 [221.8 to 437.6] | 277.5 [200.4 to 384.1]
  rSBA-MenC: number analyzed (Participants) | 51 | 63
  rSBA-MenC | 88.6 [54.2 to 144.8] | 85.5 [55.1 to 132.5]
  rSBA-MenW-135: number analyzed (Participants) | 52 | 64
  rSBA-MenW-135 | 339.4 [235.2 to 489.8] | 404.2 [308.5 to 529.7]
  rSBA-MenY | 347.6 [223.9 to 539.6] | 367.7 [287.8 to 469.9]

19. Secondary Outcome: rSBA Antibody Titers.
Description: Titers are given as geometric mean titers (GMTs), calculated for all subjects for the serogroups rSBA-MenA, rSBA-MenC, rSBAMenW-135, and rSBA-MenY respectively. Titers were determined by Public Health England (PHE) laboratory assay.
Time Frame: At Year 5 (60 months following primary vaccination)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Group Y5 | Nimenrix 2 Group Y5
Number analyzed (Participants) | 62 | 72
Titers
  rSBA-MenA: number analyzed (Participants) | 61 | 72
  rSBA-MenA | 32.4 [18.7 to 56] | 32.3 [19.1 to 54.7]
  rSBA-MenC: number analyzed (Participants) | 62 | 71
  rSBA-MenC | 20 [12 to 33.4] | 16.5 [10.2 to 26.6]
  rSBA-MenW-135 | 8.9 [5.9 to 13.6] | 11.8 [7.5 to 18.5]
  rSBA-MenY: number analyzed (Participants) | 61 | 72
  rSBA-MenY | 32 [17.8 to 57.4] | 26.9 [16.2 to 44.7]

20. Secondary Outcome: Antibody to Polysacccharide N. Meningitidis Serogroup A, C, W-135 and Y (Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY) Antibody Concentrations
Description: Results were tabulated as geometric mean antibody concentration (GMC) calculated on all subjects, expressed in microgram per milliliter (μg/ml).
Time Frame: At Year 1 (12 months post primary vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1
Number analyzed (Participants) | 103 | 120
μg/ml
  Anti-PSA | 0.45 [0.36 to 0.58] | 0.33 [0.28 to 0.4]
  Anti-PSC: number analyzed (Participants) | 102 | 114
  Anti-PSC | 0.27 [0.22 to 0.32] | 0.25 [0.22 to 0.3]
  Anti-PSW-135: number analyzed (Participants) | 99 | 113
  Anti-PSW-135 | 0.96 [0.74 to 1.25] | 1.2 [1 to 1.44]
  Anti-PSY: number analyzed (Participants) | 98 | 117
  Anti-PSY | 1.41 [1.07 to 1.85] | 1.7 [1.43 to 2.03]

21. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥ 0.3 μg/ml and ≥ 2.0 μg/ml respectively.
Time Frame: At Year 1 (12 months post primary vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Group Y1 | Nimenrix 2 Group Y1
Number analyzed (Participants) | 103 | 120
Participants
  Anti-PSA, ≥0.3 μg/ml | 60 | 59
  Anti-PSA, ≥2.0 μg/ml | 12 | 6
  Anti-PSC, ≥0.3 μg/ml: number analyzed (Participants) | 102 | 114
  Anti-PSC, ≥0.3 μg/ml | 36 | 39
  Anti-PSC, ≥2.0 μg/ml: number analyzed (Participants) | 102 | 114
  Anti-PSC, ≥2.0 μg/ml | 3 | 4
  Anti-PSW-135, ≥0.3 μg/ml: number analyzed (Participants) | 99 | 113
  Anti-PSW-135, ≥0.3 μg/ml | 78 | 104
  Anti-PSW-135, ≥2.0 μg/ml: number analyzed (Participants) | 99 | 113
  Anti-PSW-135, ≥2.0 μg/ml | 28 | 29
  Anti-PSY, ≥0.3 μg/ml: number analyzed (Participants) | 98 | 117
  Anti-PSY, ≥0.3 μg/ml | 84 | 114
  Row Anti-PSY, ≥2.0 μg/ml: number analyzed (Participants) | 98 | 117
  Row Anti-PSY, ≥2.0 μg/ml | 45 | 50

22. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titers ≥ Cut-off Values
Description: hSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off value assessed were ≥ 1:4 or 1:8. This outcome measure only concerns the Nimenrix Naive Group.
Time Frame: At Month 60 (pre-primary vaccination with Nimenrix vaccine)
Population: The analysis was performed on the Booster ATP cohort for immunogenicity,which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken before the primary vaccination with Nimenrix, of the Nimenrix Naive Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Naive Group
Number analyzed (Participants) | 79
Participants
  hSBA-MenA, ≥1:4 | 16
  hSBA-MenA, ≥1:8 | 16
  hSBA-MenC,≥1:4: number analyzed (Participants) | 71
  hSBA-MenC,≥1:4 | 28
  hSBA-MenC, ≥1:8: number analyzed (Participants) | 71
  hSBA-MenC, ≥1:8 | 24
  hSBA-MenW-135, ≥1:4: number analyzed (Participants) | 77
  hSBA-MenW-135, ≥1:4 | 28
  hSBA-MenW-135, ≥1:8: number analyzed (Participants) | 77
  hSBA-MenW-135, ≥1:8 | 28
  hSBA-MenY, ≥1:4: number analyzed (Participants) | 69
  hSBA-MenY, ≥1:4 | 29
  hSBA-MenY, ≥1:8: number analyzed (Participants) | 69
  hSBA-MenY, ≥1:8 | 29

23. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titers
Description: Titers are given as geometric mean titers (GMTs) for the serogroups hSBA-MenA, hSBA-MenC, hSBAMenW-135, and hSBA-MenY respectively. This outcome measure only concerns the Nimenrix Naive Group.
Time Frame: At Month 60 (pre-vaccination with Nimenrix vaccine)
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Naive Group
Number analyzed (Participants) | 79
Titers
  hSBA-MenA | 3.3 [2.6 to 4.1]
  hSBA-MenC: number analyzed (Participants) | 71
  hSBA-MenC | 5.3 [3.9 to 7.3]
  hSBA-MenW-135: number analyzed (Participants) | 77
  hSBA-MenW-135 | 7 [4.7 to 10.4]
  hSBA-MenY: number analyzed (Participants) | 69
  hSBA-MenY | 9.5 [5.9 to 15.1]

24. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers ≥ Cut-off Values
Description: rSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off value assessed were ≥ 1:8 or 1:128. This outcome measure only concerns the Nimenrix Naive Group.
Time Frame: At Month 60 (pre-primary vaccination with Nimenrix vaccine)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Naive Group
Number analyzed (Participants) | 78
Participants
  rSBA-MenA, ≥ 1:8 | 20
  rSBA-MenA, ≥ 1:128 | 9
  rSBA-MenC, ≥ 1:8: number analyzed (Participants) | 77
  rSBA-MenC, ≥ 1:8 | 5
  rSBA-MenC, ≥ 1:128: number analyzed (Participants) | 77
  rSBA-MenC, ≥ 1:128 | 4
  rSBA-MenW-135, ≥ 1:8 | 3
  rSBA-MenW-135, ≥ 1:128 | 3
  rSBA-MenY, ≥ 1:8 | 23
  rSBA-MenY, ≥ 1:128 | 23

25. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) for the serogroups rSBA-MenA, rSBA-MenC, rSBAMenW-135, and rSBA-MenY respectively. This outcome measure only concerns the Nimenrix Naive Group.
Time Frame: At Month 60 (pre-primary vaccination with Nimenrix vaccine)
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Naive Group
Number analyzed (Participants) | 78
Titers
  rSBA-MenA | 8.1 [5.7 to 11.5]
  rSBA-MenC: number analyzed (Participants) | 77
  rSBA-MenC | 5.2 [4.1 to 6.7]
  rSBA-MenW-135 | 4.7 [3.9 to 5.6]
  rSBA-MenY | 16.6 [9.9 to 27.7]

26. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titers ≥ Cut-off Values
Description: hSBA antibody titers were assessed for the MenA, MenC, MenW-135, and MenY serogroups respectively. The antibody cut-off values assessed were ≥ 1:4 or 1:8.
Time Frame: At Month 61, one month post-primary vaccination for Nimenrix Naive Group; one month post-booster for Nimenrix 1 and Nimenrix 2 Groups
Population: The analysis was performed on the Booster ATP cohort for immunogenicity,which included all vaccinated subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after the primary (Nimenrix Naive Group) or booster vaccination (Nimenrix1 and Nimenrix 2 Group)
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 1 Booster Group Y5: Subjects who received 1 dose on Nimenrix vaccine at 12 months of age and a booster dose of Nimenrix vaccine at Year 5 (60 months post-primary vacccination).
- Nimenrix 2 Booster Group Y5: Subjects who were previously vaccinated with two doses of Nimenrix, one each at 9 and 12 months of age and a booster dose of Nimenrix vaccine at Year 5 (60 months post-primary vacccination).
- Nimenrix Naive Group Y5: Vaccine-naive subjects aged 5-6 years were enrolled to receive Nimenrix vaccine as primary vaccination at Year 5.
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 32 | 38 | 79
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 31 | 38 | 79
  hSBA-MenA, ≥ 1:4 | 31 | 38 | 62
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 31 | 38 | 79
  hSBA-MenA, ≥ 1:8 | 31 | 38 | 62
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 32 | 37 | 77
  hSBA-MenC, ≥ 1:4 | 32 | 37 | 68
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 32 | 37 | 77
  hSBA-MenC, ≥ 1:8 | 32 | 37 | 66
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 32 | 38 | 78
  hSBA-MenW-135, ≥ 1:4 | 32 | 38 | 70
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 32 | 38 | 78
  hSBA-MenW-135, ≥ 1:8 | 32 | 38 | 70
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 32 | 38 | 70
  hSBA-MenY, ≥ 1:4 | 32 | 38 | 66
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 32 | 38 | 70
  hSBA-MenY, ≥ 1:8 | 32 | 38 | 66

27. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titers
Description: Titers were given as geometric mean titers (GMTs) for the serogroups hSBA-MenA, hSBA-MenC,hSBAMenW-135, and hSBA-MenY respectively, calculated on all subjects.
Time Frame: as for outcome 26
Population: The analysis was performed on the Booster ATP cohort for immunogenicity,which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after the primary (Nimenrix Naive Group) or booster vaccination (Nimenrix 1 and Nimenrix 2 Group)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 32 | 38 | 79
Titers
  hSBA-MenA: number analyzed (Participants) | 31 | 38 | 79
  hSBA-MenA | 1395.9 [926.0 to 2104.4] | 1590.1 [1157.4 to 2184.6] | 38.3 [25.4 to 57.9]
  hSBA-MenC: number analyzed (Participants) | 32 | 37 | 77
  hSBA-MenC | 8185.7 [4736.9 to 14145.4] | 12881.2 [8549.1 to 19408.4] | 95.3 [56.5 to 160.9]
  hSBA-MenW-135: number analyzed (Participants) | 32 | 38 | 78
  hSBA-MenW-135 | 15800.9 [12975.8 to 19241.0] | 20495.9 [16080.2 to 26124.3] | 98.1 [65.8 to 146]
  hSBA-MenY: number analyzed (Participants) | 32 | 38 | 70
  hSBA-MenY | 8809.1 [6926.3 to 11203.9] | 10513.8 [7933.6 to 13933.2] | 198.7 [137.6 to 287]

28. Secondary Outcome: Number of Subjects With Vaccine Response for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers
Description: Vaccine response was defines as: for initially seronegative subjects (pre-vaccination titer < 1:4): hSBA post-vaccination antibody titers ≥ 1:8 and for seropositive subjects (pre-vaccination titers ≥ 1:4): hSBA antibody titers at least four times the pre-vaccination antibody titers.
Time Frame: as for outcome 26
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 31 | 35 | 77
Participants
  hSBA-MenA | 31 | 35 | 56
  hSBA-MenC: number analyzed (Participants) | 30 | 34 | 68
  hSBA-MenC | 28 | 31 | 48
  hSBA-MenW-135: number analyzed (Participants) | 31 | 35 | 74
  hSBA-MenW-135 | 31 | 35 | 48
  hSBA-MenY: number analyzed (Participants) | 26 | 31 | 61
  hSBA-MenY | 26 | 31 | 48

29. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBAMenW-135 and rSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥1:8 and ≥1:128. Titers were determined by Public Health England (PHE) laboratory assay.
Time Frame: At Month 60 and 61 (just prior to and one month post-primary vaccination for Nimenrix Naive Group; one month post-booster vaccination for Nimenrix 1 and Nimenrix 2 Groups)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 31 | 38 | 82
Participants
  rSBA-MenA, M60 ≥1:8: number analyzed (Participants) | 30 | 37 | 78
  rSBA-MenA, M60 ≥1:8 | 21 | 23 | 20
  rSBA-MenA, M60 ≥1:128: number analyzed (Participants) | 30 | 37 | 78
  rSBA-MenA, M60 ≥1:128 | 11 | 14 | 9
  rSBA-MenA, M61 ≥1:8 | 31 | 38 | 81
  rSBA-MenA, M61 ≥1:128 | 31 | 38 | 81
  rSBA-MenC, M60 ≥1:8: number analyzed (Participants) | 31 | 37 | 77
  rSBA-MenC, M60 ≥1:8 | 15 | 18 | 5
  rSBA-MenC, M60 ≥1:128: number analyzed (Participants) | 31 | 37 | 77
  rSBA-MenC, M60 ≥1:128 | 6 | 12 | 4
  rSBA-MenC, M61 ≥1:8 | 31 | 38 | 80
  rSBA-MenC, M61 ≥1:128 | 31 | 38 | 72
  rSBA-MenW-135, M60 ≥1:8: number analyzed (Participants) | 31 | 37 | 78
  rSBA-MenW-135, M60 ≥1:8 | 7 | 10 | 3
  rSBA-MenW-135, M60 ≥1:128: number analyzed (Participants) | 31 | 37 | 78
  rSBA-MenW-135, M60 ≥1:128 | 4 | 7 | 3
  rSBA-MenW-135, M61 ≥1:8 | 31 | 38 | 82
  rSBA-MenW-135, M61 ≥1:128 | 31 | 38 | 81
  rSBA-MenY, M60 ≥1:8: number analyzed (Participants) | 30 | 37 | 78
  rSBA-MenY, M60 ≥1:8 | 16 | 18 | 23
  rSBA-MenY, M60 ≥1:128: number analyzed (Participants) | 30 | 37 | 78
  rSBA-MenY, M60 ≥1:128 | 10 | 12 | 23
  rSBA-MenY, M61 ≥1:8 | 31 | 38 | 82
  rSBA-MenY, M61 ≥1:128 | 31 | 38 | 82

30. Secondary Outcome: rSBA Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) for the serogroups rSBA-MenA, rSBA-MenC, rSBAMenW-135, and rSBA-MenY respectively, determined by Public Health England [PHE] laboratory assay.
Time Frame: At Month 60 and 61 (just prior to and one month post-primary vaccination for Nimenrix Naive Group; one month post-booster for Nimenrix 1 and Nimenrix 2 Groups)
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 31 | 38 | 82
Titers
  rSBA-MenA, M60: number analyzed (Participants) | 30 | 37 | 78
  rSBA-MenA, M60 | 35.9 [16.8 to 76.8] | 35.8 [17.1 to 75] | 8.1 [5.7 to 11.5]
  rSBA-MenA, M61 | 5238.1 [3835.3 to 7154.1] | 5287.7 [4212.4 to 6637.4] | 2970.7 [2282.6 to 3866.1]
  rSBA-MenC, M60: number analyzed (Participants) | 31 | 37 | 77
  rSBA-MenC, M60 | 16 [8.5 to 30] | 20 [10.1 to 39.7] | 5.2 [4.1 to 6.7]
  rSBA-MenC, M61 | 2738.9 [1707.8 to 4392.5] | 3605 [2401.2 to 5412.4] | 525.1 [365.2 to 755.2]
  rSBA-MenW-135, M60: number analyzed (Participants) | 31 | 37 | 78
  rSBA-MenW-135, M60 | 8.7 [4.9 to 15.5] | 10 [5.7 to 17.7] | 4.7 [3.9 to 5.6]
  rSBA-MenW-135, M61 | 10713.2 [7632.4 to 15037.4] | 11585.2 [8901.4 to 15078.2] | 5792.6 [4591.7 to 7307.6]
  rSBA-MenY, M60: number analyzed (Participants) | 30 | 37 | 78
  rSBA-MenY, M60 | 29.2 [12.8 to 66.3] | 22 [10.8 to 44.9] | 16.6 [9.9 to 27.7]
  rSBA-MenY, M61 | 5601.6 [4181.4 to 7504] | 5098.3 [4044.6 to 6426.5] | 4027.3 [3159 to 5134.4]

31. Secondary Outcome: Number of Subjects With Vaccine Response With rSBA-MenA, rSBA-MenC, hSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Vaccine response was defined as: for initially seronegative subjects: antibody titer ≥ 1:32 at post-vaccination; and for initially seropositive subjects: antibody titer at post-vaccination ≥ 4 fold the pre-vaccination antibody titer. Titers were determined by Public Health England (PHE) laboratory assay.
Time Frame: At Month 61 (one month post-primary vaccination for Nimenrix Naive Group; one month post-booster for Nimenrix 1 and Nimenrix 2 Groups)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 30 | 37 | 78
Participants
  rSBA-MenA: number analyzed (Participants) | 29 | 37 | 78
  rSBA-MenA | 28 | 36 | 75
  rSBA-MenC: number analyzed (Participants) | 30 | 37 | 77
  rSBA-MenC | 26 | 32 | 70
  rSBA-MenW-135 | 30 | 37 | 77
  rSBA-MenY: number analyzed (Participants) | 29 | 37 | 78
  rSBA-MenY | 29 | 36 | 78

32. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptom
Description: Assessed solicited local symptoms were pain, redness and swelling. Any was defined as occurrence of the symptom regardless of intensity grade. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness/swelling was defined as redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-primary vaccination for Nimenrix Naive Group and post-booster for Nimenrix 1 and Nimenrix 2 Groups
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in this current study who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 36 | 45 | 89
Participants
  Any Pain | 18 | 21 | 46
  Grade 3 Pain | 0 | 1 | 1
  Any Redness | 10 | 15 | 22
  Grade 3 Redness | 1 | 0 | 1
  Any Swelling | 8 | 9 | 21
  Grade 3 Swelling | 1 | 0 | 2

33. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptom
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache and gastrointestinal. Any was defined as occurrence of the symptom regardless of their intensity grade or relationship to study vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever higher than (>) 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 36 | 45 | 89
Participants
  Any Fatigue | 10 | 7 | 18
  Grade 3 Fatigue | 0 | 0 | 1
  Related Fatigue | 8 | 6 | 15
  Any Gastrointestinal | 4 | 5 | 7
  Grade 3 Gastrointestinal | 1 | 2 | 0
  Related Gastrointestinal | 3 | 4 | 5
  Any Headache | 4 | 5 | 11
  Grade 3 Headache | 1 | 1 | 1
  Related Headache | 4 | 4 | 8
  Any Fever (Axillary) | 1 | 2 | 5
  Fever (Axillary) >39.5°C | 0 | 0 | 0
  Related Fever (Axillary) | 0 | 1 | 3

34. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-primary vaccination for Nimenrix Naive Group and post-booster for Nimenrix 1 and Nimenrix 2 Groups
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in this current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 38 | 46 | 100
Participants | 9 | 6 | 29

35. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the 181-day (Days 0-180) post primary vaccination for Nimenrix Naive Group and post booster for Nimenrix 1 and Nimenrix 2 Groups
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 38 | 46 | 100
Participants | 0 | 0 | 1

36. Secondary Outcome: Number of Subjects Reporting Any New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: as for outcome 35
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1 Booster Group Y5 | Nimenrix 2 Booster Group Y5 | Nimenrix Naive Group Y5
Number analyzed (Participants) | 38 | 46 | 100
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period; Unsolicited adverse events (AEs): during the 31-day (Days 0-30) post-vaccination period; Serious adverse events (SAEs): during the entire study period (from Day 0 up to Month 54).
Description: Unsolicitied AEs and SAEs were assessed on the Total Vaccinated Cohort. Solicited symptoms were assessed on those subjects from the Total Vaccinated Cohort who returned their symptom sheet.
Arm/Group | Nimenrix 1 Group | Nimenrix 2 Group | Nimenrix Naive Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/46 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/46 | 1/100
Other Adverse Events (participants affected / at risk) | 31/38 | 43/46 | 67/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix 1 Group (N=38) | Nimenrix 2 Group (N=46) | Nimenrix Naive Group (N=100)
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix 1 Group (N=38) | Nimenrix 2 Group (N=46) | Nimenrix Naive Group (N=100)
Pain (General disorders) | 18/36 | 21/45 | 46/89
Redness (General disorders) | 10/36 | 15/45 | 22/89
Swelling (General disorders) | 8/36 | 9/45 | 21/89
Fatigue (General disorders) | 10/36 | 7/45 | 18/89
Gastrointestinal symptoms (General disorders) | 4/36 | 5/45 | 7/89
Headache (General disorders) | 4/36 | 5/45 | 11/89
Fever (General disorders) | 1/36 | 2/45 | 5/89
Injection site bruising (Injury, poisoning and procedural complications) | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.